CLINICAL TRIAL: NCT00006241
Title: A Pivotal Study to Determine the Safety and Efficacy of Using B-Cell High Density Microparticles (BCell-HDM) to Deplete B-Cells From Peripheral Blood Stem Cell Collections Without Compromising the Time to Neutrophil and Platelet Engraftment in Patients With Relapsed Low or Intermediate Grade B-Cell Non-Hodgkin's Lymphoma Given Autologous Peripheral Blood Stem Cell Transplants After High-Dose Chemotherapy
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Relapsed Low- or Intermediate-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1488.00; FHCRC-1488.00; ELIGIX-C99-105; NCI-G00-1846; CDR0000068166 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-09-11; First posted 2004-06-22 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Drug Therapy; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: chemotherapy
Procedure: in vitro-treated peripheral blood stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy. Treating the peripheral stem cells in the laboratory to remove any existing cancer cells may improve the effectiveness of the transplant.

PURPOSE: Randomized phase II trial to compare the effectiveness of treated peripheral stem cells with that of untreated stem cells in patients who have relapsed low- or intermediate-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effectiveness of the B-cell high density microparticles (BCell-HDM) device in purging B-cells from peripheral blood stem cells (PBSC) harvested from patients with relapsed low or intermediate grade B-cell non-Hodgkin's lymphoma. II. Determine the recovery of T-cells and CD34+ cells in BCell-HDM processed PBSC in these patients. III. Compare hematopoietic engraftment following infusion of autologous PBSC purged using the BCell-HDM device versus unpurged autologous PBSC in these patients receiving high dose chemotherapy. IV. Determine the toxicity of this regimen in these patients. V. Determine the occurrence of adverse effects from this regimen in these patients.

OUTLINE: This is a randomized, double blind, multicenter study. Patients are stratified by grade of lymphoma (low vs intermediate), type of myeloablative conditioning regimen (chemotherapy only vs chemotherapy/total body irradiation), and center. Patients are randomized to one of two treatment arms. Patients undergo peripheral blood stem cell (PBSC) harvest over no more than 4 consecutive days. A myeloablative conditioning regimen of either chemotherapy alone or chemotherapy/total body irradiation is given within 4 weeks of PBSC harvest. Prior to randomization one patient at each center receives PBSC transplantation using cells purged with the B-cell high density microparticle (BCell-HDM) device. Arm I: Patients receive BCell-HDM treated PBSC transplantation on day 0. Arm II: Patients receive untreated PBSC transplantation on day 0. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 1 and continuing until blood counts recover. Patients are followed on days 30 and 100, and then at 6 and 12 months.

PROJECTED ACCRUAL: A total of 115 patients (15 for prerandomization study, 50 for each treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of relapsed low or intermediate grade B-cell non-Hodgkin's lymphoma CD20+ or CD19+ tumor cells Bone marrow involvement less than 20% of intratrabecular space All tumor masses less than 5 cm in each dimension In second or greater remission with either complete remission or minimal disease state OR Failed to achieve remission with primary induction therapy, but can achieve minimal disease with additional chemotherapy or radiotherapy OR Persistent splenomegaly with otherwise minimal disease No active CNS involvement A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: LVEF at least 45% Pulmonary: DLCO at least 50% predicted Other: Not pregnant Negative pregnancy test No prior other malignancy except carcinoma in situ of the cervix or basal cell carcinoma of the skin No known hypersensitivity to nickel No known hypersensitivity to mouse proteins HIV negative HTLV I and II negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since prior unconjugated anti-B-cell monoclonal antibody (mAb) (e.g., rituximab, Campath I) No prior anti-B-cell mAb conjugated to radioisotopes such as iodine I 131 (e.g., iodine I monoclonal antibody anti-B1) or yttrium Y No concurrent mAb therapy until 12 months after study No other biologic therapy (e.g., monoclonal antibodies, interferon alfa) for 12 months after study No concurrent hematopoietic growth factors other than filgrastim (G-CSF) Chemotherapy: See Disease Characteristics No chemotherapy within 5 days prior to PBSC collection No other concurrent chemotherapy for 12 months after study Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No concurrent radiotherapy for 12 months after study Surgery: Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03; Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States